CLINICAL TRIAL: NCT00088049
Title: A Randomized Double-Blind Study of Olanzapine Versus Aripiprazole in the Treatment of Schizophrenia
Brief Title: Study of Olanzapine vs. Aripiprazole in the Treatment of Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8047; F1D-MC-HGLB
Record Dates: First submitted 2004-07-19; First posted 2004-07-21 (Estimated); Last update posted 2007-07-18 (Estimated); Status verified 2007-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine; Aripiprazole

INTERVENTIONS:
Drug: Olanzapine
Drug: Aripiprazole

SUMMARY:
The purpose of the protocol is to evaluate the efficacy of olanzapine compared with Aripiprazole in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female inpatient or outpatients, ages 18-65

Exclusion Criteria:

* Participation in a clinical trial of another drug including olanzapine or aripiprazole within 30 days prior to study entry (visit 1).
* Treatment with clozapine within the past 12 months.
* Have known uncorrected narrow-angle glaucoma.
* Have a diagnosis of Parkinson's disease, dementia or related disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560
Dates: Start 2003-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To determine the long-term effectiveness and tolerability as measured by time to all-cause treatment discontinuation of olanzapine and aripiprazole relative to each other in patients with schizophrenia during 28 weeks of double-blind therapy

SECONDARY OUTCOMES:
To assess olanzapine versus aripiprazole in the following:
improvement in psychopathology of schizophrenia as measured by PANSS change
change in CGI-S and PGI-I scores
level of activation as measured by PANSS change
depressive symptoms as measured by MADRS score
response rates
time to failure to maintain response
quality of life as measured by the SWN-S and SF-36
cognitive functioning as measured by the MOS
sexual functioning as measured by the GISF
health resource utilization and resource utilization costs
hospitalization time
treatment emergent adverse events
EPS as measured by the Simpson-Angus, Barnes, and AIMS
laboratory values
vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (24):
- United States (24):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Garden Grove, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, National City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Oakbrook Terrace, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Glen Burnie, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Cedarhurst, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Scranton, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Salt Lake City, Utah

REFERENCES:
- [Derived] Liu-Seifert H, Ascher-Svanum H, Osuntokun O, Jen KY, Gomez JC. Change in level of productivity in the treatment of schizophrenia with olanzapine or other antipsychotics. BMC Psychiatry. 2011 May 17;11:87. doi: 10.1186/1471-244X-11-87. PMID 21586165
- [Derived] Ascher-Svanum H, Stensland MD, Peng X, Faries DE, Stauffer VL, Osuntokun OO, Kane JM. Cost-effectiveness of olanzapine vs. aripiprazole in the treatment of schizophrenia. Curr Med Res Opin. 2011 Jan;27(1):115-22. doi: 10.1185/03007995.2010.537594. Epub 2010 Nov 26. PMID 21110749
- [Derived] Kane JM, Osuntokun O, Kryzhanovskaya LA, Xu W, Stauffer VL, Watson SB, Breier A. A 28-week, randomized, double-blind study of olanzapine versus aripiprazole in the treatment of schizophrenia. J Clin Psychiatry. 2009 Apr;70(4):572-81. doi: 10.4088/jcp.08m04421. Epub 2009 Mar 24. PMID 19323965